CLINICAL TRIAL: NCT05945914
Title: Oncoplastic Entirely Robot-Assisted Approach (OPERA) - Incorporating Robotic Surgery in Both Mastectomy and DIEP Flap Reconstruction
Brief Title: Incorporating Robotic Surgery in Both Mastectomy and DIEP Flap Reconstruction
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Ju Huang, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202300888B0
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with unilateral breast cancer received robotic-assisted mastectomy and robotic assisted free DIEP flap harvest for breast reconstruction.
  Interventions: Procedure: Oncoplastic Entirely Robot-Assisted Approach (OPERA)

INTERVENTIONS:
Procedure: Oncoplastic Entirely Robot-Assisted Approach (OPERA) — Robotic-assisted surgery in both mastectomy and free DIEP flap harvest, so-called Oncoplastic Entirely Robot-Assisted Approach (OPERA).

SUMMARY:
A prospective study will be conducted to assess the outcomes of patients who underwent concurrent robotic-assisted mastectomy and robotic-assisted free DIEP flap harvest for breast reconstruction between March 2020 and June 25, 2023. Demographic data, including age, body mass index (BMI), and medical history, were collected, along with surgical time and perioperative parameters. The incidence of acute and chronic complications was documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral breast cancer received robotic-assisted mastectomy and robotic assisted free DIEP flap harvest for breast reconstruction

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unilateral breast cancer received robotic-assisted mastectomy and robotic assisted free DIEP flap harvest for breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Re-open | Post-operative 14 days
  Whether the patient return to the operation room to check the blood flow or re-do the anastomosis.
Acute complication (< 30 days) | Post-operative 30 days
Chronic complication (> 30 days) | One year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan